CLINICAL TRIAL: NCT03181230
Title: Pilot Study of Health, Fitness, and Quality of Life in Adolescent Girls With Turner Syndrome
Brief Title: Health, Fitness, and Quality of Life in Adolescent Girls With Turner Syndrome
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0142; UL1TR001082 (NIH)
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Turner Syndrome; Turner Syndrome Mosaicism, 45, X/46, XX or XY; Turner Syndrome Mosaicism 46,X,I(X)(Q10)/45,X; Turner Syndrome Karyotype 46,X With Abnormal Sex Chromosome , Except I(Xq)
Keywords: Turner syndrome; 45,XO; body composition; cardiometabolism; quality of life; fitness
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents: Adolescents and young adults with Turner syndrome will undergo studies of cardiometabolism, fitness, quality of life questionnaires, and a brief interview.
  Interventions: Other: No intervention
- Parents: One parent of a participant will complete parent-report quality of life questionnaires and a brief interview.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study plans to learn more about how the energy system works in girls with Turner syndrome. This is important to know so that the investigators understand how Turner syndrome relates to diseases such as diabetes, extra weight gain, heart disease and liver disease, and how this impacts day to day life.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12-21 years
* 45,XO karyotype in >50% of cells tested with a diagnosis of Turner syndrome (TS)
* Tanner stage 2-5 for breast development

Exclusion Criteria:

* Growth hormone treatment within the past 3 months
* Diagnosis of type 1 or type 2 diabetes
* Untreated hypertension with blood pressure > 99%ile for sex, age and height or >140/90
* Weight > 300 lbs
* Height < 54"
* Aortic sinus of Valsalva or ascending aorta z-score > 2
* Other cognitive, psychiatric, or physical impairment resulting in inability to tolerate the study procedures, including vigorous exercise
* Pregnancy

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Investigators will enroll adolescent and young adult females with Turner syndrome who will complete all study procedures. One parent will also be enrolled (either mother or father) to complete questionnaires about the daughter.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | Baseline
  Peak oxygen consumption (VO2 peak) with a standard graded exercise (bicycle) test

SECONDARY OUTCOMES:
Quality of Life Survey | Baseline
  Self and parent reported quality of life
Percent body fat | Baseline
  Body composition by dual-energy x-ray absorptiometry
Insulin resistance (IR) | Baseline
  Fasting insulin and glucose used to calculate homeostatic model assessment (HOMA)

OTHER OUTCOMES:
Qualitative structured interview | Baseline
  Attitudes surrounding physical activity participation

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee Davis, MD, MS, Principal Investigator — University of Colroado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No